CLINICAL TRIAL: NCT04823832
Title: Endoscopic Versus Percutaneous Biliary Drainage for Resectable Pancreatic Head Cancer With Hyperbilirubinemia and Impact on Pancreaticoduodenectomy: A Prospective Cohort Study
Brief Title: Endoscopic Versus Percutaneous Biliary Drainage for Resectable Pancreatic Head Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hani Alhadad (Other)
Responsible Party: Sponsor-Investigator, Hani Alhadad, assistant professor, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30/11
Record Dates: First submitted 2021-02-23; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Head Cancer; Obstructive Jaundice
MeSH Terms: conditions — Jaundice, Obstructive | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERCP group (Active Comparator): endoscopic retrograde cholangiopancreaticography with plastic stent insertion
  Interventions: Procedure: pancreaticoduodenectomy
- PTD group (Active Comparator): ultrasound guided percutaneous transhepatic catheter insertion
  Interventions: Procedure: pancreaticoduodenectomy

INTERVENTIONS:
Procedure: pancreaticoduodenectomy — resection of the head of pancreas and the duodenum followed by triple anastomosis
  Other Names: whipple operation

SUMMARY:
Patients with potentially resectable pancreatic head cancer and high bilirubin level, were stratified into two equal groups according to the method of biliary drainage: endoscopic stenting or percutaneous drainage.

DETAILED DESCRIPTION:
Along with history taking and complete clinical examination, the results of complete blood count, international normalized ratio , renal and liver function tests were obtained. Patients with coagulopathy were corrected by fresh frozen plasma and repeated vitamin K injections to reach an INR of at least 1.4 before the intervention, otherwise, they were excluded. Besides, ultrasound and computed tomography of the abdomen/pelvis (pancreatic protocol) were routinely undertaken. Tumors were staged for resectability according to TNM staging system.

Patients were randomly divided by closed envelope method into two groups; patients were allocated to the first group (ERCP) who underwent Endoscopic Retrograde Cholangio-Pancreatography coupled with placement of a 10-French plastic stent; and to the second group (PTD) who underwent Fluoroscopy-guided Percutaneous Transhepatic Drainage.

Preoperative biliary drainage Parenteral broad spectrum antibiotics were administered prior and after each intervention. ERCP was performed under general anesthesia in the operation room and a 10-french (3.2 mm) covered polyethylene stent with side flaps to prevent migration was placed below the level of biliary bifurcation. Stents were inserted over a guidewire via an Olympus 4.2 mm channel endoscope, by standard techniques.

PTD was placed in the interventional radiology department under local anesthesia via the left duct sub-xiphoid approach, only via the external approach. A 6 french gauge catheter was positioned with its tip above the biliary obstruction. After PTD, patients were instructed to drink a lot of fluids to replace fluid loss or they were given temporary intravenous fluid supplementation.

After either procedure, patients were either discharged home or kept in hospital. Those who were discharged were readmitted for preoperative preparation. Patients were followed up clinically as well as by laboratory results. The total and direct bilirubin level and other liver function tests were repeated after ten days from the procedure to estimate the decline in their levels. Post-intervention complications either PTD-related such as bleeding, cholangitis, bile leak and catheter occlusion/displacement; or ERCP-related such as pancreatitis, cholangitis, bleeding and stent displacement; were recorded.

Surgery After improvement of liver functions, patients were scheduled for PD. All operations were performed through a hockey-stick incision by consultant surgeons experienced in pancreatic surgery. The standard surgical procedure was pancreaticoduodenectomy with pylorus preservation. The effects of pre-operative drainage were evaluated during the operation in terms of operative resection time, blood loss, difficulties of dissection and intra-operative bleeding. While the endoscopic stent is removed intra-operatively after transection of the common hepatic duct, the catheter of PTD is left and inserted in the hepaticojejunostomy (stented anastomosis) to be removed two weeks later. Perioperative complications (< 30 days) were stratified for each group according to Clavien-Dindo classification.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant obstruction of the distal common bile duct e.g. adenocarcinoma of the pancreatic head or periampullary tumor
* Hyperbilirubinemia, total bilirubin level more than 10 mg/dL
* Cholangitis, pruritis, coagulopathy, nausea and anorexia

Exclusion Criteria:

* Patients with advanced disease
* metastatic disease
* Patients undergoing neoadjuvant therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
number of participants with operative difficulties as assessed by the operating surgeon | up to 6 hours at the time of surgery
  measuring the difficulty of dissection, number of operative complications encountered
number of participants with post operative complications | up to one month
  detection of postoperative complications in the early postoperative period

SECONDARY OUTCOMES:
number of participants with postprocedural complications | up to one month after each procedure
  detection of postprocedure complications

CONTACTS AND LOCATIONS:
Overall Officials: Wael N Abdelsalam, doctor, Study Director — dean of faculty
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
to keep the confidentiality of each patient

DOCUMENTS (2):
  • Study Protocol (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT04823832/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT04823832/SAP_001.pdf